CLINICAL TRIAL: NCT05214755
Title: Translation, Cross-Cultural Adaptation and Turkish Validation of the 25-Question Geriatric Locomotive Function Scale
Status: Completed | Type: Observational
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, Büşra Aksan Sadıkoğlu, Physiotherapist, Istanbul Aydın University
Other Study IDs: IstanbulAU2022
Record Dates: First submitted 2022-01-17; First posted 2022-01-31 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Translation, Cultural Adaptation and Turkish Validation
Keywords: Elderly; Turkish; GLFS-25; Function; Reliability; Validity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
25-question Geriatric Locomotive Function Scale (GLFS-25) is a patient-reported outcome measure consisting of 25 questions that evaluates locomotive functions and locomotive syndrome risk in elderly individuals.

The purpose of this study was to translate and cross-culturally adapt the English version of the GLFS-25 into Turkish and to investigate the reliability and validity of the translated version of the scale.

DETAILED DESCRIPTION:
Aging is an inevitable process that begins after birth and continues until the death of the individual, affecting the person mentally and physically. Approximately 21% of elderly individuals requiring care have locomotive organ disorders involving the bone, joint, muscle and nervous system. 25-question Geriatric Locomotive Function Scale (GLFS-25), developed by Japanese researchers in 2012, is a patient-reported outcome measure consisting of 25 questions that evaluates locomotive functions and locomotive syndrome risk in elderly individuals. This scale provides an advantage in terms of locomotive ability and early detection of locomotive syndrome in the elderly. In addition, the scale provides the opportunity to decrease number of needing for hospital care of elderly individuals by early detection of locomotive functions and the risk of locomotive syndrome. Before a patient-reported outcome measure can be used in a society other than the one in which it was developed, it must be translated and culturally adapted. The GLFS-25 have been translated to different cultural settings and into many languages, including Brazilian, Iranian and Chinese. Data obtained from the culturally adapted versions contribute to a better understanding of the tools measurement properties. The studies reported that translated versions of GLFS-25 reliable and valid in older adults for functional assessment. Therefore, a Turkish version of the GLFS-25 would likely be that would be helpful in the functional state management and risk factor analyzes for locomotive syndrome of the Turkish older adult population. The purpose of this study was to translate and cross-culturally adapt the English version of the GLFS-25 into Turkish and to investigate the reliability and validity of the translated version of the scale.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 65
* who can answer the questionnaire on their own or with the help of their relatives

Exclusion Criteria:

* unable to walk without the assistance of another person
* having a brain disease or severe cardiovascular, pulmonary or renal disease
* having a history of lower extremity and/or spine fractures in the last 6 months
* were treated for acute trauma

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — over the age of 65 (Older Adult)
Study Population: Elderly people who are over the age of 65 and can answer the questionnaire on their own or with the help of their relatives.
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
25-question Geriatric Locomotive Function Scale (GLFS-25) | Baseline
  GLFS-25 is an assessment tool developed for evaluate locomotive functions in elderly individuals. This scale consists of a self-reported questionnaire with 25 items that are easily understood by the elderly, and each item is graded from 0 to 4 points. The final score is determined by the sum of all items ranging from 0 to 100.

SECONDARY OUTCOMES:
25-question Geriatric Locomotive Function Scale (GLFS-25) | Within a 7-to-14-day period after the first assessment
  GLFS-25 is an assessment tool developed for evaluate locomotive functions in elderly individuals. This scale consists of a self-reported questionnaire with 25 items that are easily understood by the elderly, and each item is graded from 0 to 4 points. The final score is determined by the sum of all items ranging from 0 to 100.
Katz Index | Baseline
  The scale consists of 6 questions evaluating washing, dressing, toilet, continence, transfer and feeding activities. For activities, 'dependent' is evaluated with 0 point and 'independent' is evaluated with 1 point. Six points indicate complete independence, 0 point complete dependence.
Lawton Index | Baseline
  This index includes 8 activities: the ability to use a phone, shopping, using public transport, meal preparation, doing daily housework, traveling, the responsibility for using medication and the ability to handle finance. The scoring scale is 0 and 1, and the sum of the scores is varied from 0 to 8 points.
Visual Analogue Scale (VAS) | Baseline
  The VAS assesses pain status on a 10 cm chart, with 0 points defined as "no pain" and 10 points as "terrible pain".
Geriatric Depression Scale | Baseline
  Geriatric Depression Scale is a 30-item scale that evaluates the level of depression in elderly individuals. Questions 1,5,7,9,15,19,21,28,29 and 30 in the scale are evaluated with 0 point for 'yes' and 1 point for 'no'. The total scoring is 30 points, and individuals who score 14 are reported to have a high risk of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrrahpasa, Istanbul, Turkey (Türkiye)